CLINICAL TRIAL: NCT07114731
Title: The Comparison of the Effects of Synchronous and Asynchronous Action Observation Therapy on Balance, Walking and Functional Capacity in Children With Cerebral Palsy
Brief Title: Comparison of Synchronous and Asynchronous Action Observation Therapy in Children With Cerebral Palsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Iremnur Gunhan, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulUC_IG
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy (CP); Spastic Diplegia Cerebral Palsy; Spastic Hemiplegic Cerebral Palsy; Neurodevelopmental Disorder (Diagnosis); Action Observation; Action Observation Therapy
Keywords: Pediatric Rehabilitation; Neurodevelopmental Disorders; Cerebral Palsy; Action Observation Therapy; Neuroplasticity; Motor Learning; Children; Mirror Neuron System; Motor Function
MeSH Terms: conditions — Cerebral Palsy; Cerebral palsy, spastic, diplegic; Neurodevelopmental Disorders; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodevelopmental treatment (NDT) + Synchronous Action Observation Therapy (AOT) Group (Experimental): Participants in this group will receive a 20-minute Neurodevelopmental Training (NDT) session followed by synchronous Action Observation Therapy (AOT). The AOT component consists of four video modules:
  1. Sitting position + Sit-to-Stand exercises
  2. Weight-shifting exercises
  3. Balance exercises
  4. Walking exercises
  Participants will observe the videos in real-time and perform the movements simultaneously. The intervention will last for 8 weeks, with sessions conducted twice weekly for 45 minutes each.
  Interventions: Other: Synchronous Action Observation Therapy
- Neurodevelopmental treatment (NDT) + Asynchronous Action Observation Therapy (AOT) Group (Experimental): Participants in this group will receive the same 20-minute NDT session followed by asynchronous Action Observation Therapy (AOT). In this group, participants will first watch each of the four video modules, then perform the exercises afterward (i.e., not in real time).
  The intervention will last for 8 weeks, with sessions conducted twice weekly for 45 minutes each.
  Interventions: Other: Asynchronous Action Observation Therapy

INTERVENTIONS:
Other: Synchronous Action Observation Therapy — Real-time observation and execution of motor tasks through structured video modules designed based on participants' GMFCS level and extremity involvement.
  Arms: Neurodevelopmental treatment (NDT) + Synchronous Action Observation Therapy (AOT) Group
Other: Asynchronous Action Observation Therapy — Observation of structured motor task videos followed by delayed execution, adapted to individual GMFCS levels and extremity involvement patterns.
  Arms: Neurodevelopmental treatment (NDT) + Asynchronous Action Observation Therapy (AOT) Group

SUMMARY:
The aim of this study is to compare the effects of synchronous and asynchronous action observation therapy (AOT) on balance, gait, and functional capacity in children with cerebral palsy (CP). CP is a neurodevelopmental disorder characterized by impairments in motor skills, particularly motor control and postural balance. By examining the contributions of synchronous (real-time) and asynchronous (delayed) AOT methods to motor performance, this study seeks to identify the most effective therapeutic approach for this population.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is defined as a non-progressive neurological disorder that arises during fetal development, the neonatal period, or early childhood and results in permanent motor impairments. Lesions in the central nervous system of children with CP lead to a range of musculoskeletal, neuromuscular, and sensory system problems, causing postural abnormalities, balance and coordination deficits, and limitations in mobility. These impairments significantly reduce independence in activities of daily living.

Various therapeutic approaches are utilized in the rehabilitation process to improve the functional independence of children with CP. According to the International Classification of Functioning, Disability and Health (ICF), rehabilitation interventions should be grounded in neuroplasticity-based principles to maximize functional outcomes. One such neuroplasticity-based approach that has gained increasing attention in recent years is Action Observation Therapy (AOT).

AOT is based on the mirror neuron theory, which posits that observing an action activates similar neural regions in the cerebral cortex as performing the action itself. This simultaneous activation facilitates action understanding, imitation, and motor learning, suggesting that AOT may be an effective intervention to enhance motor function in individuals with CP. Improving motor functions in children with CP is crucial to enhancing their participation in daily life activities and overall quality of life. In addition to conventional physiotherapy interventions, AOT has emerged in recent years as an effective rehabilitation strategy that supports neuroplasticity. AOT facilitates motor learning and skill acquisition by targeting the brain's mirror neuron system.

Although there is substantial evidence in the literature demonstrating that AOT improves upper extremity functions, studies systematically comparing its effects on balance, gait, and general functional capacity remain limited. In particular, the differential effects of synchronous and asynchronous AOT applications on various motor outcomes have not yet been thoroughly investigated. Understanding the mechanisms of action of these two approaches may contribute to the development of more individualized and tailored treatment programs for children with CP.

Moreover, the low cost and easy applicability of AOT increase its potential for clinical use. Therefore, the findings of this study could enhance the effectiveness of rehabilitation programs, offering more accessible treatment alternatives for both healthcare professionals and families. To address this gap in the literature, the present study aims to comprehensively investigate the effects of synchronous and asynchronous AOT on motor functions in children with CP.

In this study, both groups will receive neurodevelopmental treatment (NDT) for 20 minutes as part of their intervention program. In addition, participants in the synchronous AOT group will observe exercise videos divided into four components (1. Sitting posture and sit-to-stand exercises; 2. Weight-shifting exercises; 3. Balance exercises; 4. Gait exercises) and perform the observed movements simultaneously in real time. Conversely, the asynchronous AOT group will first observe each of these video segments for 3 minutes and then perform the corresponding exercises sequentially after observation. Each session will last 45 minutes, conducted twice a week for 8 weeks.

The exercise videos were developed to include 12 task-oriented exercises tailored to the GMFCS level and extremity involvement of the children. The exercises are designed with varying levels of difficulty to enhance functional skills and lower extremity performance.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation of both the child and their family in the study
* Diagnosis of cerebral palsy with spastic clinical type, including hemiparetic and diparetic distribution
* Age between 6 and 18 years
* Classified as Level I or II according to the Gross Motor Function Classification System (GMFCS)
* Ability to comply with exercise interventions (based on medical report indicating normal mental level or "mild mental retardation")
* Ability to understand and speak Turkish

Exclusion Criteria:

* Presence of spasticity ≥3 in lower extremity muscle groups as measured by the Modified Ashworth Scale
* Inability to cooperate with verbal commands
* Presence of visual or hearing impairments
* Diagnosis of epilepsy or current use of antiepileptic medications
* Presence of joint contractures
* Botulinum toxin injection to the lower extremities within the past 6 months
* Undergoing orthopedic surgery within the past 6 months
* Presence of any additional systemic or neurological diseases
* Missing three consecutive rehabilitation sessions

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure - 88 (GMFM-88) - Dimensions D and E | 2 days before treatment and 8 weeks
  The GMFM-88 is a standardized observational instrument designed to measure changes in gross motor function in children with cerebral palsy. The scale consists of five dimensions:
  (A) Lying and rolling
  (B) Sitting
  (C) Crawling and kneeling
  (D) Standing
  (E) Walking, running, and jumping
  For this study, only Dimensions D and E will be assessed to evaluate standing and locomotor abilities. Each item is scored based on the child's ability to perform specific motor tasks. Scores can be calculated for each dimension separately as well as combined for a total score.
Pediatric Balance Scale (PBS) | 2 days before treatment and 8 weeks
  The pediatric balance scale is a modified version of the Berg balance scale and is used to evaluate the functional balance ability of school-age children. The scale consists of 14 items, scored from 0 (lowest function) to 4 (highest function), with a maximum score of 56.

SECONDARY OUTCOMES:
Gross Motor Function Classification System | 2 days before treatment
  The Gross Motor Function Classification System (KMFSS) for CP is based on self-initiated movements with an emphasis on sitting, displacement and mobility. The main criterion when defining the five-level classification system is that the differences between the levels are meaningful in everyday life.
  General titles of each level LEVEL I: Walks without restrictions. LEVEL II: Walks with restrictions. LEVEL III: Walks using hand-held mobility devices. LEVEL IV: Self-movement is limited. Can use a motorized mobility vehicle. LEVEL V: Transported in a manual wheelchair.
Gillette Functional Assessment Questionnaire (FAQ) | 2 days before treatment and 8 weeks
  The FAQ is a parent-reported tool designed to assess functional walking ability in children. It evaluates the level of independence and mobility in various daily walking activities, providing a global rating of walking performance.
10-Meter Walk Test (10MWT) | 2 days before treatment and 8 weeks
  The 10MWT is a timed performance test used to assess walking speed over a short distance. Participants are asked to walk a 10-meter path at their usual pace, and the time (in seconds) is recorded. The test is commonly used in pediatric populations with mobility limitations.
Five Times Sit to Stand Test | 2 days before treatment and 8 weeks
  This test evaluates lower extremity functional strength and transitional movements. Participants are instructed to stand up and sit down five times consecutively as fast as possible from a standard chair without using their arms. The total time to complete the task is recorded.
Functional Reach Test (FRT) | 2 days before treatment and 8 weeks
  The FRT assesses dynamic balance by measuring the maximal distance a participant can reach forward and sideways while standing in a fixed position without losing balance. A tape measure is mounted at shoulder height on the wall to track the reach distance.
Timed Get Up and Go Test (TUG) | 2 days before treatment and 8 weeks
  It is a valid and reliable method used to evaluate functional mobility and static and dynamic balance in CP. From a starting position with hips, knees, and ankles flexed to 90°, participants get up from a chair without arm support, walk 3 meters, return and sit in the chair. The time starts to be recorded with the "go" prompt given by the evaluator and is stopped when the hip touches the chair.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Unıversıty-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided